CLINICAL TRIAL: NCT06701734
Title: Targeted Translocator Protein PET Imaging Evaluate Neuroinflammation of the Chronic Pain Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Weibing Miao, PhD (Other)
Responsible Party: Sponsor-Investigator, Weibing Miao, PhD, professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: Chronic_pain_DPA714 PET
Record Dates: First submitted 2024-11-16; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Chroinc Pain; PET; Microglial Activation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Chronic pain is a major public health issue, which seriously affects patients' quality of life. Neuroinflammation is an important mechanism resulting in chronic pain. Translocator protein (TSPO) has served as a marker of microglial activation and neuroinflammation. 18F-DPA714, a tracer targeted TSPO, can be used to evaluate the microglial activation and neuroinflammation in vivo by PET imaging.Recent and increasing studies have found changes in TSPO and its ligands in various chronic pain models. Reversing their expressions has been shown to alleviate chronic pain in these models, illustrating the effects of TSPO and its ligands.The investigators aim to explore the clinical feasibility used 18F-DPA714 PET imaging to monitor microglial cells activation of center nervous system in chronic pain patients. This study might reveal significant neuroinflammatory process in the center nervous system of the chronic pain patients. The results of this study might provide a new biomarker of disease pathological progression and indicates that TSPO-based therapy may become an alternative strategy for treating chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain patients
* Written informed consent was provided by the patients and their family

Exclusion Criteria:

* history of head trauma ， epilepsy， claustrophobia, rheumatic or autoimmune diseases, psychiatric disorders, severe somatic diseases (neurological,cardiovascular, etc.),previous heart or brain surgery, substance abuse, inability to refrain from hypnotics, magnetic implants, pregnancy, lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Value | 2 years
  Measures of specific binding of 18F-DPA-714 measures of specific binding of the tracer